CLINICAL TRIAL: NCT02973152
Title: Does Laryngeal Reinnervation or Type I Thyroplasty Give Better Voice Results for Patients With Unilateral Vocal Fold Paralysis (VOCALIST): a Feasibility Study.
Brief Title: Laryngeal Reinnervation Versus Thyroplasty in Patients With Vocal Fold Weakness.
Acronym: VOCALIST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal National Throat, Nose and Ear Hospital (Other)
Collaborators: University College Joint Research Office (Unknown); University College London Hospitals (Other); National Institute for Health Research, United Kingdom (Other Government); Sealed Envelope: Redpill Online Application (Unknown)
Responsible Party: Principal Investigator, Professor Martin Birchall, Professor, Royal National Throat, Nose and Ear Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11/0107; PB-PG-1013-32058 (Other: University College London Hospitals NHS Foundation Trust)
Record Dates: First submitted 2016-11-03; First posted 2016-11-25 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Vocal Cord Paralysis Unilateral
Keywords: Type I Thyroplasty; Reinnervation
MeSH Terms: conditions — Vocal Cord Paralysis | interventions — Laryngoplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thyroplasty (Active Comparator): This medialisation/augmentation technique is a static technique, performed under local anaesthesia that aims to improve the positioning of the paralysed vocal fold. It uses a silastic implant readily available in different sizes according to size of larynx and gender of the patient. The correct size can be determined intraoperatively by using a measuring device while listening and visualising the larynx with flexible fiberoptic scope simultaneously.
  Interventions: Procedure: Thyroplasty
- Reinnervation (Active Comparator): For laryngeal reinnervation, ansa cervicalis to recurrent laryngeal nerve repair technique will be used. In this technique, the functioning ansa cervicalis nerve that overlies the internal jugular vein and the distal stump of injured recurrent laryngeal nerve (RLN) will be identified and anastomosed without tension (Crumley RL. Teflon versus thyroplasty versus nerve transfer: a comparison. The Annals of otology, rhinology, and laryngology. 1990;99(10 Pt 1):759-63).
  Interventions: Procedure: Reinnervation

INTERVENTIONS:
Procedure: Thyroplasty — This medialisation/augmentation technique is a static technique, performed under local anaesthesia that aims to improve the positioning of the paralysed vocal fold. It uses a silastic implant readily available in different sizes according to size of larynx and gender of the patient. The correct size can be determined intraoperatively by using a measuring device while listening and visualising the larynx with flexible fiberoptic scope simultaneously.
  Arms: Thyroplasty
Procedure: Reinnervation — For laryngeal reinnervation, ansa cervicalis to recurrent laryngeal nerve repair technique will be used. In this technique, the functioning ansa cervicalis nerve that overlies the internal jugular vein and the distal stump of injured recurrent laryngeal nerve (RLN) will be identified and anastomosed without tension (Crumley RL. Teflon versus thyroplasty versus nerve transfer: a comparison. The Annals of otology, rhinology, and laryngology. 1990;99(10 Pt 1):759-63).
  Arms: Reinnervation

SUMMARY:
The purpose of this study is to help determine the most effective treatment for participants with Unilateral Vocal Fold Paralysis.

There are currently two types of operations used to treat this condition. One operation is called thyroplasty. Doctors place a small piece of safe plastic into the side of the participant's voice box to push the weak vocal cord into a position to enable better speech and swallowing. In the other operation called laryngeal reinnervation, doctors repair the neck nerve supply to the vocal cord using parts of other unaffected nerves to enable better speech and swallowing. The investigators do not know which of these methods is better and are conducting this study to start comparing the two operations so that a larger clinical trial can be conducted in the future to tell us which operation is best.

DETAILED DESCRIPTION:
Title: Does Laryngeal Reinnervation or Type I Thyroplasty give better voice results for patients with Unilateral Vocal Fold Paralysis (VOCALIST): a feasibility study

Short title: VOCALIST

Trial medication: Not Applicable

Phase of trial: Phase IIb

Objectives: The aim of the study is to establish the feasibility of a multicentre, randomised phase III clinical trial of surgical treatment for Unilateral Vocal Fold Paralysis (UVFP).

Main objectives are to test the feasibility of:

1. the multicentre recruitment process, including continuous improvement to the process based on qualitative analysis;
2. recruiters being able to present true equipoise with the treatment arms;
3. the randomisation process and investigate reasons for any difficulties that affect recruitment
4. the utility of the following characteristics of the proposed primary (voice handicap index) and secondary outcomes: variability across patients, variability over time, differences in outcome between randomised groups over time;
5. process of follow up visits and diary completion;
6. means of gathering health economics and health-related quality of life data suitable for measuring cost effectiveness.

Type of trial: Quantitative and Qualitative Feasibility Study; multi-centre randomised controlled trial

Trial design and methods: 30 patients will be randomised to receive the Laryngeal Reinnervation or Type I Thyroplasty surgery.

Trial duration per participant: 12 months

Estimated total trial duration: 24 months

Planned trial sites: Multi-site; London, Poole and Manchester (3 sites).

Total number of participants planned: 30

Statistical methodology and analysis: The trial analysis will be descriptive and will be performed on an intention to treat basis. Primary and secondary outcomes will be described using proportions and means as appropriate, with confidence intervals. No formal comparisons will be made. The correlations between the voice outcome measures will be calculated. There is no planned interim analysis.

ELIGIBILITY:
Inclusion Criteria:

* UVFP due to unilateral recurrent laryngeal nerve paralysis of traumatic, iatrogenic or idiopathic origin of between 6 and 60 months duration. Or symptoms that have not sufficiently improved with speech therapy alone, as determined by the patient and agreed by a multidisciplinary clinical team, after 6 months and pending a surgical decision.
* Age from 18 to 70 years old
* Male or female
* Able to provide informed consent
* A significant voice disorder as measured by perceptual rating (Grade ≥2 GRBAS Scale) and Voice Handicap Index (VHI-10 score >16)
* Common laryngeal electromyography (EMG, neurophysiological) criteria (Koufman Grades 2-5) in either the thyroarytenoid (TA) or posterior cricoarytenoid (PCA) muscle on the paralysed side.

Exclusion Criteria:

* Impaired vocal fold mobility but a normal EMG (Koufman Grade I)
* Severe lung disorders
* Structural vocal fold lesions such as polyp
* Previous laryngeal framework surgery
* Cricoarytenoid joint fixation (CAJF)
* Significant non-laryngeal speech abnormality (severe dysarthria determined by a panel of trained speech therapists)
* Previous Level 2, 3 or 4 thyroid neck dissection
* Previous ipsilateral surgical neck dissection
* Previous radiotherapy to the head and neck
* Laryngeal injection of a rapidly absorbable material in the last 6 months.
* Previous laryngeal injection of a non-rapidly absorbable material (e.g. bioplastics, VOX)
* Neuromuscular disease affecting the larynx or multiple cranial nerve palsies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-05; Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Whether the participant was randomised (yes/no) | 24 months
  From those participants who were eligible to enter the study, whether the participant was randomised (yes/no)
Whether the participant successfully received the allocated operation (yes/no) | 24 months
  From those participants who were eligible to enter the study, whether the participant successfully received the allocated operation (yes/no)
Whether the participant completed the trial (yes/no) | 24 months
  From those participants who were eligible to enter the study, whether the participant completed the trial (yes/no)

SECONDARY OUTCOMES:
Whether the Study Management Group (SMG) and recruiters are in clinical equipoise in relation to treatment arms (yes/no) measured by Qualitative researcher via interviews. | 24 months
  Assessed by a Qualitative researcher via interviews with SMG members/recruiters which will explore views on the trial design and treatment groups ('arms'), perceptions of uncertainty/equipoise, views about eligibility criteria, and accounts of how the protocol is delivered in practice.
Whether surgeons and speech therapists are in clinical equipoise in relation to treatment arms (yes/no) measured by Qualitative researcher via interviews. between the two treatments | 24 months
  Assessed by a Qualitative researcher via interviews with SMG members/recruiters which will explore views on the trial design and treatment groups ('arms'), perceptions of uncertainty/equipoise, views about eligibility criteria, and accounts of how the protocol is delivered in practice.
Patient views and beliefs on randomisation, recruitment and retention measured by Qualitative researcher via interviews. processes | 24 months
  Assessed by a Qualitative researcher via interviews with patients will explore the acceptability of the trial interventions and trial processes and reasons for participation / non-participation (where applicable).
Patient and surgeon/speech therapist views on utility of chosen outcome measure measured by Qualitative researcher via interviews. measures | 24 months
  Assessed by a Qualitative researcher via interviews with SMG members/recruiters which will explore views on the trial design and treatment groups ('arms'), perceptions of uncertainty/equipoise, views about eligibility criteria, and accounts of how the protocol is delivered in practice. Interviews with patients will explore the acceptability of the trial interventions and trial processes and reasons for participation / non-participation (where applicable).
Interaction between recruiter and patient during recruitment process measured by Qualitative researcher via interviews. | 24 months
  Assessed by a Qualitative researcher via interviews with SMG members/recruiters which will explore views on the trial design and treatment groups ('arms'), perceptions of uncertainty/equipoise, views about eligibility criteria, and accounts of how the protocol is delivered in practice.Interviews with patients will explore the acceptability of the trial interventions and trial processes and reasons for participation / non-participation (where applicable).
The validated EQ-5D-5L questionnaire will be used to evaluate the participants' health-related quality of life | Baseline, 6 months and 12 month post surgery
  The secondary outcome measures will be plotted against time, and outcome differences between the surgical groups will be estimated, with 95% confidence intervals, using ANCOVA methodology that adjusts for baseline outcome measures.
The validated VHI-10 [134] will be used to evaluate the psychosocial effects of voice disorder. | Baseline, 6 months and 12 month post surgery
  The secondary outcome measures will be plotted against time, and outcome differences between the surgical groups will be estimated, with 95% confidence intervals, using ANCOVA methodology that adjusts for baseline outcome measures.
The validated Eating Assessment Tool (EAT-10) [1920] will be used to evaluate the effects of swallowing. | Baseline, 6 months and 12 month post surgery
  The secondary outcome measures will be plotted against time, and outcome differences between the surgical groups will be estimated, with 95% confidence intervals, using ANCOVA methodology that adjusts for baseline outcome measures.
The Stroboscopy Research Instrument (SRI) scale will be used to rate the Vocal cord vibration. | Baseline, 6 months and 12 month post surgery
  The secondary outcome measures will be plotted against time, and outcome differences between the surgical groups will be estimated, with 95% confidence intervals, using ANCOVA methodology that adjusts for baseline outcome measures.
Perceptual voice quality analysis will be determined using the GRBAS scale. | Baseline, 6 months and 12 month post surgery
  The secondary outcome measures will be plotted against time, and outcome differences between the surgical groups will be estimated, with 95% confidence intervals, using ANCOVA methodology that adjusts for baseline outcome measures.
The OperaVOX™ system will also be used to perform the acoustic voice analysis. | Baseline, 6 months and 12 month post surgery
  The secondary outcome measures will be plotted against time, and outcome differences between the surgical groups will be estimated, with 95% confidence intervals, using ANCOVA methodology that adjusts for baseline outcome measures.
The validated 100ml Water Swallow test will be used to measure the participants' swallowing. | Baseline, 6 months and 12 month post surgery
  The secondary outcome measures will be plotted against time, and outcome differences between the surgical groups will be estimated, with 95% confidence intervals, using ANCOVA methodology that adjusts for baseline outcome measures.
Laryngeal EMG will be used to detect laryngeal muscle activity. | Baseline, 6 months and 12 month post surgery
  The secondary outcome measures will be plotted against time, and outcome differences between the surgical groups will be estimated, with 95% confidence intervals, using ANCOVA methodology that adjusts for baseline outcome measures.
Cost of laryngeal reinnervation versus thyroplasty procedures for unilateral vocal fold paralysis. | 24 months
  A detailed cost analysis of laryngeal reinnervation and thyroplasty procedures will be undertaken, since these are likely to be major cost components affecting the relative cost-effectiveness of laryngeal reinnervation. This will include the costs of the index procedure (staff costs, theatre costs, costs of consumables, recovery costs), length of hospital stay for index procedure, post-operative ibuprofen, and speech and language therapy. Costs for the index procedure will be obtained from the hospital finance department.
Lifetime incremental cost per quality-adjusted life year QALY gained of laryngeal reinnervation versus thyroplasty. | 24 months
  An analysis of the feasibility study for a full economic evaluation of laryngeal reinnervation versus thyroplasty that will accompany the Phase III trial. This will be based on the idea that we will be aiming estimate the lifetime incremental cost per quality-adjusted life year (QALY) gained of laryngeal reinnervation versus thyroplasty, the outcome measure recommended by NICE when evaluating the cost-effectiveness of health care programmes in the NHS.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Martin Birchall, FRCS,FMedSci, Principal Investigator — University College London Hospitals
Locations (1):
- Royal National Throat Nose and Ear Hospital, 330 Gray's Inn Road, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided